CLINICAL TRIAL: NCT03443492
Title: A Phase II Randomized Study of SLOG vs mFOLFIRINOX as the First-line Treatment in Locally Advanced Uncresectable or Metastatic Pancreatic Cancer
Brief Title: SLOG vs mFOLFIRINOX as the First-line Treatment in Locally Advanced Uncresectable or Metastatic Pancreatic Cancer
Acronym: Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University (Other); Taipei Medical University Shuang Ho Hospital (Other); Chang Gung Memorial Hospital (Other); Tri-Service General Hospital (Other); E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T5217
Record Dates: First submitted 2018-02-08; First posted 2018-02-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2019-11

CONDITIONS: Locally Advanced or Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); Gemcitabine; Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLOG (Experimental): 800 mg/m2 gemcitabine at a fixed rate of 10 mg/m2/min followed by a 2-hour intravenous infusion of oxaliplatin on day 1 plus twice daily oral S-1 80-120 mg/day (based on BSA) and oral leucovorin 30 mg twice a day on day 1 to day 7, every 14 days as a cycle
  Interventions: Drug: S-1; Drug: Leucovorin(oral ); Drug: Gemcitabine; Drug: Oxaliplatin
- mFOLFIRINOX (Experimental): oxaliplatin at a dose of 85 mg/m2, given as a 2-hour infusion, with the addition, after 30 minutes, of irinotecan at a dose of 150 mg/m2, given as a 90-minute infusion. The treatment was immediately followed by a continuous intravenous infusion via central venous catheter of leucovorin 400 mg/m2 given as a 2-hour infusion and 5-FU 2400 mg/m2 over a 46-hour period on day 1 every 14 days/cycle.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: 5-FU; Drug: Leucovorin(IV)

INTERVENTIONS:
Drug: S-1 — Intervention is administered to patients in this Arm.
  Arms: SLOG
Drug: Leucovorin(oral ) — Intervention is administered to patients in this Arm.
  Arms: SLOG
Drug: Gemcitabine — Intervention is administered to patients in this Arm.
  Arms: SLOG
Drug: Oxaliplatin — Intervention is administered to patients in this Arm.
Drug: Irinotecan — Intervention is administered to patients in this Arm.
  Arms: mFOLFIRINOX
Drug: 5-FU — Intervention is administered to patients in this Arm.
  Arms: mFOLFIRINOX
Drug: Leucovorin(IV) — Intervention is administered to patients in this Arm.
  Arms: mFOLFIRINOX

SUMMARY:
A randomized phase II study to compare the efficacy and safety of SLOG or mFOLFIRINOX as a first-line treatment for patients with locally advanced and metastatic pancreatic cancer.

DETAILED DESCRIPTION:
A total 130 patients (65 patients per arm) with locally advanced or metastatic pancreatic cancer will be enrolled in multiple hospitals of Taiwan. The primary endpoint is progression-free survival. The secondary endpoints are objective response rate, overall survival and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have cyto-/histologically confirmed, locally advanced unresectable or metastatic adenocarcinoma of the pancreas (mPAC). Patients who have disease measurable or evaluable on x-ray, CT scan, or physical examination are eligible.
2. Patients must have no history of prior chemotherapy for PAC, except those delivered as adjuvant setting that completed at least 6 months before documentation of recurrence by imaging study.
3. Patients with prior radiotherapy are eligible if the irradiated area does not involve the only source of measurable / evaluable disease.
4. Patients' baseline ECOG performance status must be 1.
5. Patients' life expectancy 12 weeks or greater.
6. Patients' age 20 and 80.
7. Patients with biliary obstruction and adequate drainage procedures before enrollment are eligible.
8. Patients must agree to have indwelling venous catheter implanted.
9. Women or men and their partners of reproductive potential should agree to use an effective contraceptive method.
10. All patients must be informed of the investigational nature of this study and must sign and give written informed consent.

Exclusion Criteria:

1. Patients who have major abdominal surgery, radiotherapy or other investigating agents within 4 weeks are not eligible. Patients who have palliative radiotherapy for bony metastasis will be eligible 2 weeks after the completion of radiotherapy.
2. Patients with central nervous system metastasis
3. Patients with active infection
4. Pregnant or breast-nursing women
5. Patients with active cardiopulmonary disease or history of ischemic heart disease
6. Patients who have peripheral neuropathy > Grade I of any etiology
7. Patients who have serious concomitant systemic disorders incompatible with the study, i.e. poorly controlled diabetes mellitus, auto-immune disorders, cirrhosis of the liver, and the rest will be at the discretion of in-charged investigator.
8. Patients who have other prior or concurrent malignancy except for adequately treated in situ carcinoma of cervix or adequately treated basal cell carcinoma of skin, or any malignancy remains disease-free for 3 or more years after initial curative treatment
9. Patients who are under biologic treatment for their malignancy
10. Laboratory tests (hematology, chemistry) outside specified limits:

    1. WBC ≤ 3 x 10³/mm³
    2. ANC ≤ 1.5 x 10³/mm³
    3. Platelets ≤ 100.000/mm³
    4. Hb ≤ 9.0 g/dl (≤ 5.6 mmol/l)
    5. GFR < 60 mL/min
    6. AST and/or ALT > 2.5 x ULN; for patients with significant liver metastasis AST and/or ALT > 5 x ULN
    7. Total bilirubin > 2 x ULN
    8. Albumin < 2.5 g/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
progression free survival (PFS) | Since this is an exploratory trial, it takes a sample size of 61 patients per arm entered in 2 years with a minimum 1 year of follow up to reach 75% power with type I error of 10% under the assumptions of exponential survival functions.
  The 6-month PFS rates of the two arms are assumed to be 60% (SLOG) vs. 45% (mFOLFIRINOX)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Li-Tzong, Study Chair — National Insitute of Cancer Research
Locations (1):
- National Institute of Cancer Research, Miaoli, Taiwan

REFERENCES:
- [Derived] Chiang NJ, Tsai KK, Hsiao CF, Yang SH, Hsiao HH, Shen WC, Hsu C, Lin YL, Chen JS, Shan YS, Chen LT. A multicenter, phase I/II trial of biweekly S-1, leucovorin, oxaliplatin and gemcitabine in metastatic pancreatic adenocarcinoma-TCOG T1211 study. Eur J Cancer. 2020 Jan;124:123-130. doi: 10.1016/j.ejca.2019.10.023. Epub 2019 Nov 22. PMID 31765987